CLINICAL TRIAL: NCT02753283
Title: Sustaining Skeletal Health in Frail Elderly
Brief Title: Preventing Osteoporosis Using Denosumab
Acronym: PROUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Susan L. Greenspan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Susan L. Greenspan, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY19050268; 1R01AG052123-01 (NIH)
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis; Osteoporotic Fractures
Keywords: Bone loss; Frail Geriatric Patients; Nursing Home Patients; Long-term Care Patients; Osteoporosis; Osteoporotic Fractures
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Osteoporotic Fractures; Bone Diseases, Metabolic | interventions — Denosumab; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Women Denosumab (Experimental): Semi-annual dose for women: denosumab 60 mg semi-annual injection; Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplements).
  Interventions: Drug: denosumab; Dietary Supplement: Calcium and Vitamin D
- Women Placebo Group (Placebo Comparator): Semi-annual for women: placebo saline injection; Vitamin D 800-1000 IU/daily and Calcium approximately1200 mg/daily (dietary + supplements).
  Interventions: Drug: Placebo; Dietary Supplement: Calcium and Vitamin D
- Men Denosumab (Experimental): Semi-annual dose for men: denosumab 60 mg semi-annual injection; Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplements).
  Interventions: Drug: denosumab; Dietary Supplement: Calcium and Vitamin D
- Men Placebo Group (Placebo Comparator): Semi-annual for men: placebo saline injection; Vitamin D 800-1000 IU/daily and Calcium approximately1200 mg/daily (dietary + supplements)
  Interventions: Drug: Placebo; Dietary Supplement: Calcium and Vitamin D

INTERVENTIONS:
Drug: denosumab — Semi-annual dose: 60 mg injection; Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplement)
  Other Names: Prolia
  Arms: Men Denosumab; Women Denosumab
Drug: Placebo — Semi-annual saline injection
  Arms: Men Placebo Group; Women Placebo Group
Dietary Supplement: Calcium and Vitamin D — Dietary supplement: Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplement)

SUMMARY:
The purpose of this research study is to find out if denosumab (Prolia®), an injection given in the arm under the skin every 6 months, works to treat bone loss and prevent it from worsening in older men and women (ages 65 and older) who have osteoporosis and reside in long-term care (LTC) facilities.

DETAILED DESCRIPTION:
Objective:

The long term goal is to improve health, well-being and quality of life in the frail long-term care (LTC) elderly population by reducing fractures. The short term goal is to demonstrate efficacy of the non-bisphosphonate denosumab to improve bone mineral density (BMD), a necessary (but not sufficient) pre-condition of a large fracture reduction trial. The investigators propose to conduct a 2-year, randomized, double-blind, calcium-vitamin D controlled trial to test the efficacy and predictability of the antiresorptive RANK ligand inhibitor, denosumab (60 mg), among a cohort of 212 institutionalized, under-served, frail men and women ≥65 years old in LTC.

Specific Aims:

Aim 1: To evaluate efficacy of denosumab in improving/maintaining bone mineral density. The investigators will measure conventional hip and spine bone mineral density (BMD).

Primary Hypothesis: After 2 years, women and men on denosumab will have greater hip and spine BMD increases.

ELIGIBILITY:
Inclusion Criteria:

Ambulatory male and female residents with osteoporosis or low bone mass (at risk for fracture) ages 65 and older will be considered if:

* Reside in long-term care institution (nursing home or assisted living facility); and
* HaveOsteoporosis: (1) by bone density [spine, hip or forearm Bone Mineral Density (BMD) T-score ≤ -2.5]; (2) A previous adult fragility fracture of the spine or hip; or (3) Would be treated based on FRAX® and the National Osteoporosis Foundation (NOF) treatment thresholds of a 10 year risk of ≥ 20% for a major fracture or ≥ 3% for hip fracture suing femoral neck BMD.

Exclusion Criteria:

* Institutionalized residents with subacute illnesses who are not expected to survive or who will be discharged in < 2 years.
* Non-ambulatory residents (those who cannot stand and pivot with assistance in order to transfer to the DXA table).
* Those currently on therapy (including bisphosphonate, denosumab, or teriparatide) or who have been on a bisphosphonate for > 1year during the previous 2 years because some bisphosphonates are long acting.
* Those with a history of hypocalcemia or contraindication for treatment. We will screen for these conditions by detailed history, chart review, and baseline laboratory analyses.
* Those with vitamin D levels < 25ng/mL will be treated with vitamin D 50,000 IU/wk for 8 weeks; they will be enrolled if the follow-up vitamin D level is 25 ng/mL or more (if after 2 rounds of vitamin D repletion their vitamin D level is not at least 25 ng/mL, they will not be eligible to be randomized into the study).
* Those on dialysis or with stage 5 chronic kidney disease (eGFR<15ml/min) will be excluded at screening.
* Those requiring tooth extraction or oral surgery will not be enrolled until cleared by a dentist.
* Patients will be allowed to continue on glucocorticoids and anticonvulsants because their use is common in this population.
* Those on glucocorticoids and anticonvulsants will be allowed to continue in the study because their use is common in this population.
* Those on hormone replacement therapy (HRT), raloxifene, or prescribed protective hip pads by their Primary Care Physician (PCP) will be allowed to participate and continue on these therapies.
* We will suggest that participants stop long-term calcitonin as it has been discontinued in Europe due to cancer concerns.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Greenspan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Senior Communities, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group
Started | 62 | 61 | 40 | 38
Completed | 45 | 43 | 28 | 27
Not Completed | 17 | 18 | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group | Total
Number analyzed (Participants) | 62 | 61 | 40 | 38 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 81.5 (7.6) | 80.0 (9.0) | 82.6 (8.9) | 82.7 (7.6) | 81.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 0 | 0 | 123
  Male | 0 | 0 | 40 | 38 | 78
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 4 | 6 | 1 | 1 | 12
  White | 58 | 55 | 37 | 37 | 187
  Other | 0 | 0 | 2 | 0 | 2
Bone Density of the Hip [Mean (Standard Deviation); unit: g/cm^2] | .783 (.114) | .748 (.142) | .923 (.163) | .884 (.143) | .821 (.154)
Bone Density of Spine [Mean (Standard Deviation); unit: g/cm^2] | 1.038 (.178) | 1.044 (.187) | 1.221 (.217) | 1.204 (.205) | 1.108 (.210)

OUTCOME MEASURES:

1. Primary Outcome: Bone Density of the Total Hip
Description: Bone Mineral Density (BMD) of the total hip percent change over 24 months as assessed by dual-energy x-ray absorptiometry (DXA)
Time Frame: 24 months
Measure: Mean (Standard Error); unit: Percent change
Groups:
- Men Denosumab: Semi-annual dose for women: denosumab 60 mg semi-annual injection; Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplements).
  denosumab: Semi-annual dose: 60 mg injection; Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplement)
  Calcium and Vitamin D: Dietary supplement: Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplement)
- Men Placebo Group: Semi-annual for Women: placebo saline injection; Vitamin D 800-1000 IU/daily and Calcium approximately1200 mg/daily (dietary + supplements).
  Placebo: Semi-annual saline injection
  Calcium and Vitamin D: Dietary supplement: Vitamin D 800-1000 IU/daily and Calcium approximately 1200 mg/daily (dietary + supplement)
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group
Number analyzed (Participants) | 40 | 38 | 24 | 24
Percent change | 4.62 (0.62) | -0.19 (0.79) | 3.74 (0.55) | 0.48 (0.74)
Statistical Analysis 1: Comparison: Women Denosumab vs Women Placebo Group; Test type: Superiority; p = .007, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = 4.80, Standard Error of Mean 1.48
Statistical Analysis 2: Comparison: Men Denosumab vs Men Placebo Group; Test type: Superiority; p = .018, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = 2.70, Standard Error of Mean 1.09

2. Primary Outcome: Bone Density of the Spine
Description: Bone Mineral Density (BMD) of the spine percent change over 24 months as assessed by dual-energy x-ray absorptiometry (DXA)
Time Frame: 24 months
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group
Number analyzed (Participants) | 42 | 41 | 26 | 25
Percent change | 7.41 (0.93) | 2.15 (0.56) | 7.91 (0.96) | 1.12 (1.13)
Statistical Analysis 1: Comparison: Women Denosumab vs Women Placebo Group; Test type: Superiority; p = .014, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = 3.99, Standard Error of Mean 1.45
Statistical Analysis 2: Comparison: Men Denosumab vs Men Placebo Group; Test type: Superiority; p = .002, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = 5.16, Standard Error of Mean 1.45

3. Secondary Outcome: Distal Radius BMD
Description: Percent change over 24 months
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group
Number analyzed (Participants) | 43 | 40 | 26 | 25
Percent change from baseline | 2.030 (3.322) | -.376 (3.894) | 2.386 (4.187) | -1.115 (3.455)
Statistical Analysis 1: Comparison: Women Denosumab vs Women Placebo Group; Test type: Superiority; p = .060, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = 2.54, Standard Error of Mean 1.26
Statistical Analysis 2: Comparison: Men Denosumab vs Men Placebo Group; Test type: Superiority; p = .055, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = 2.45, Standard Error of Mean 1.22

4. Secondary Outcome: Femoral Neck BMD
Description: Percent change over 24 months
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group
Number analyzed (Participants) | 40 | 38 | 24 | 24
Percent change from baseline | 3.212 (5.207) | .185 (4.195) | 2.932 (3.574) | -.958 (5.926)
Statistical Analysis 1: Comparison: Women Denosumab vs Women Placebo Group; Test type: Superiority; p = .112, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = 2.21, Standard Error of Mean 1.37
Statistical Analysis 2: Comparison: Men Denosumab vs Men Placebo Group; Test type: Superiority; p = .070, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = 2.46, Standard Error of Mean 1.34

5. Secondary Outcome: TBS
Description: Trabecular Bone Score (TBS) Percent change over 24 months. This not a scale. Higher values are better.
Time Frame: 24 Months
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group
Number analyzed (Participants) | 36 | 37 | 22 | 20
Percent change from baseline | 3.007 (5.990) | 1.099 (5.498) | 2.370 (6.645) | 3.318 (6.688)
Statistical Analysis 1: Comparison: Women Denosumab vs Women Placebo Group; Test type: Superiority; p = .904, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = -.17, Standard Error of Mean 1.39
Statistical Analysis 2: Comparison: Men Denosumab vs Men Placebo Group; Test type: Superiority; p = .616, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = -1.17, Standard Error of Mean 2.29

6. Other Pre Specified Outcome: CTX
Description: Bone Turnover Marker change from Baseline
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group
Number analyzed (Participants) | 47 | 42 | 35 | 29
nmol/L | -.190 (.206) | -.078 (.181) | -.178 (.211) | -.071 (.177)
Statistical Analysis 1: Comparison: Women Denosumab vs Women Placebo Group; Test type: Superiority; p < .001, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = -.16, Standard Error of Mean .04
Statistical Analysis 2: Comparison: Men Denosumab vs Men Placebo Group; Test type: Superiority; p = .005, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = -.09, Standard Error of Mean .03

7. Other Pre Specified Outcome: P1NP
Description: Bone Turnover Marker Change from Baseline
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group
Number analyzed (Participants) | 47 | 42 | 35 | 29
ug/L | -25.345 (21.367) | -3.158 (22.633) | -19.539 (28.219) | -10.731 (21.548)
Statistical Analysis 1: Comparison: Women Denosumab vs Women Placebo Group; Test type: Superiority; p = .001, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = -26.2, Standard Error of Mean 6.0
Statistical Analysis 2: Comparison: Men Denosumab vs Men Placebo Group; Test type: Superiority; p = .038, Mixed Models Analysis; Using multiple imputation for missing data; Mean Difference (Final Values) = -8.2, Standard Error of Mean 3.9

ADVERSE EVENTS:
Time Frame: 24 Months
Description: Subjects were asked every six months about adverse events, supplemented by automated reporting system
Arm/Group | Women Denosumab | Women Placebo Group | Men Denosumab | Men Placebo Group
All-Cause Mortality (participants affected / at risk) | 1/62 | 4/61 | 4/40 | 2/38
Serious Adverse Events (participants affected / at risk) | 21/62 | 26/61 | 21/40 | 15/38
Other Adverse Events (participants affected / at risk) | 46/62 | 50/61 | 32/40 | 33/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Women Denosumab (N=62) | Women Placebo Group (N=61) | Men Denosumab (N=40) | Men Placebo Group (N=38)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 3 | 4 | 2
Chest Pain (Cardiac disorders) | 1 | 4 | 1 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Dry Eye (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small bowel obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Complication associated with device (General disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 4 | 4 | 2
Incarcerated hernia (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0
Bacteremia (Infections and infestations) | 2 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Ankle fracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Femur Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hip fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Inflammatory polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rib fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Adenosquamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 0 | 0
Confusional state (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Internal capsule infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Ischemic cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Normal Pressure Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 1
Transient ischemic attack (Nervous system disorders) | 3 | 0 | 1 | 0
Device malfunction (Product Issues) | 0 | 1 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Genitourinary tract infection (Renal and urinary disorders) | 1 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 2 | 3 | 0 | 0
Urosepsis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Adenoviral upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Lobar Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Aortic valve replacement (Surgical and medical procedures) | 0 | 0 | 1 | 0
Brachytherapy to prostate (Surgical and medical procedures) | 0 | 0 | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 3 | 0 | 1
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 2 | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Embolic stroke (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Women Denosumab (N=62) | Women Placebo Group (N=61) | Men Denosumab (N=40) | Men Placebo Group (N=38)
Diarrhea (Gastrointestinal disorders) | 4 | 2 | 1 | 1
Fatigue (General disorders) | 1 | 0 | 3 | 0
Pain (General disorders) | 0 | 1 | 2 | 0
Bronchitis (Infections and infestations) | 3 | 2 | 2 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 2 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 4 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 24 | 24 | 16 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 9 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2 | 2
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 1
Confusional State (Nervous system disorders) | 0 | 1 | 3 | 0
Dizziness (Nervous system disorders) | 3 | 1 | 3 | 1
Headache (Nervous system disorders) | 3 | 1 | 0 | 3
Syncope (Nervous system disorders) | 0 | 1 | 2 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 1 | 3
Urinary Tract Infection (Renal and urinary disorders) | 7 | 8 | 2 | 2
Adenoviral Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 1
Skin Infection (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT02753283/Prot_SAP_000.pdf